CLINICAL TRIAL: NCT00891657
Title: A Randomised, Prospective, Multi-Centre Clinical Study of SprayShield™ Adhesion Barrier System as a Barrier for the Prevention of Adhesion Formation After Laparoscopic Myomectomy
Brief Title: Post Market Study for an Adhesion Barrier Following Laparoscopic Myomectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GYN-08-002
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Results first posted 2010-08-31 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-08

CONDITIONS: Fibroid; Myoma; Leiomyoma
Keywords: Adhesion; Fibroid; Myoma; Leiomyoma; Myomectomy
MeSH Terms: conditions — Leiomyoma; Myoma; Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SprayShield™ (Experimental): SprayShield™
  Interventions: Device: SprayShield™
- Control (No Intervention): No adhesion barrier administered.

INTERVENTIONS:
Device: SprayShield™ — Anti-adhesion barrier
  Arms: SprayShield™

SUMMARY:
This study is planned as a prospective, randomised, parallel, controlled, multi-centre, open label, comparative evaluation of SprayShield™ Adhesion Barrier plus good surgical technique, versus good surgical technique alone, with a blinded, third party video evaluation of adhesion formation at second look laparoscopy (SLL) following laparoscopic myomectomy.

ELIGIBILITY:
Inclusion Criteria:

* Females, 18 years of age or older, of child-bearing potential.
* Subject has at least one myoma >= 3 cm.

Exclusion Criteria:

* Pregnant or lactating females.
* Females undergoing prior open or closed myomectomy for treatment of myomas.
* Evidence of current active endometriosis or infection
* History of or active inflammatory bowel disease or pelvic inflammatory disease.
* Presence of a frozen pelvis, or hydrosalpinges.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rudy Leon De Wilde, MD, Principal Investigator — Pius Clinic
Locations (1):
- Pius Clinic, Oldenburg, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 10, 2008 and March 4, 2009, a total of 15 subjects were consented for potential participation, of whom all 15 subjects were randomized. There were no intra-operative screen failures.
Groups:
- SprayShield™: The SprayShield™ is a synthetic, sprayable polyethylene glycol (PEG) based absorbable gel adhesion barrier, that consists of two liquids that when mixed together rapidly cross-link to form a biocompatible absorbable flexible hydrogel that conforms and adheres to the tissues to which it is applied.
- Control: The subjects randomized to the Control group received standard good surgical care, excluding any use of anti-adhesion products.
Period: Overall Study
Arm/Group | SprayShield™ | Control
Started | 9 | 6
Completed | 8 | 5
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SprayShield™ | Control | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (4.6) | 44.3 (3.3) | 39.2 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Sites Adherent to the Uterus
Description: The number of times an adhesion is attached to the uterus.
Time Frame: 8-12 weeks post myomectomy
Population: Number of subjects to have had a second laparoscopic look.
Measure: Mean (Standard Deviation); unit: Adhesion Sites
Arm/Group | SprayShield™ | Control
Number analyzed (Participants) | 8 | 5
Adhesion Sites | 1.1 (1.0) | 0.6 (0.9)

2. Primary Outcome: Mean Severity Score of Sites Adherent to the Uterus
Description: The scoring for severity is as follows: 0=no adhesions, 1=filmy, avascular adhesions, 2=vascular and/or dense adhesions, and 3=cohesive adhesions.
Time Frame: 8-12 weeks post myomectomy
Population: Number of subjects to have had a second laparoscopic look.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | SprayShield™ | Control
Number analyzed (Participants) | 8 | 5
Scores on a Scale | 1.63 (1.06) | 0.8 (1.1)

3. Primary Outcome: Mean Extent Score of Sites Adherent to the Uterus
Description: 0 =no adhesions, 1=covering <25% of locations' total area, 2=covering 26% to 50% of locations' total area, and 3=covering >51% of locations' total area.
Time Frame: 8-12 weeks post myomectomy
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | SprayShield™ | Control
Number analyzed (Participants) | 8 | 5
Scores on a Scale | 0.92 (0.66) | 0.6 (0.89)

4. Primary Outcome: Area of Sites Adherent to the Uterus (cm^2)
Time Frame: 8-12 weeks post myomectomy
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | SprayShield™ | Control
Number analyzed (Participants) | 8 | 5
cm^2 | 2.19 (2.32) | 2.7 (5.24)

ADVERSE EVENTS:
Time Frame: 10 November 2008 (first subject consented) to 09 May 2009 (last subject follow-up visit date)
Arm/Group | SprayShield™ | Control
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/6
Other Adverse Events (participants affected / at risk) | 0/9 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SprayShield™ (N=9) | Control (N=6)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The very small sample size makes it difficult to detect any real differences between the treatments, if such differences exist.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No